CLINICAL TRIAL: NCT04898231
Title: Multisystem Inflammatory Syndrome Therapies in Children (MISTIC) Comparative Effectiveness Study
Brief Title: MIS-C Comparative Effectiveness Study
Acronym: MISTIC
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: Children's Hospital of Michigan (Other)
Responsible Party: Principal Investigator, Adriana H. Tremoulet, Associate Director, Kawasaki Disease Research Center Professor of Pediatrics, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202109
Record Dates: First submitted 2021-05-13; First posted 2021-05-24 (Actual); Results first posted 2025-11-04 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-10

CONDITIONS: Multisystem Inflammatory Syndrome-Children
MeSH Terms: interventions — Infliximab; CT-P13; Interleukin 1 Receptor Antagonist Protein; Methylprednisolone

STUDY DESIGN:
Intervention Model Description: This is a randomized trial of 3 treatment arms
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Infliximab (Active Comparator): Infliximab will be administered as a single IV dose of 10 mg/kg over 2 hours.
  Interventions: Drug: Infliximab
- Methylprednisilone (steroids) (Active Comparator): Methylprednisilone (steroids) will be administered as 2 mg/kg IV or orally divided every 12 hours. At the time of hospital discharge the patient will be given a steroid taper that will take at least 3 weeks to complete.
  Interventions: Drug: Methylprednisolone
- Anakinra (Active Comparator): Anakinra will be administered at a dose of 8 mg/kg/day IV or SQ with 100 mg every 6 hours as the max dose. This is discontinued with a taper during the hospitalization over 2-4 days once a patient is stable with significantly improved clinical course and laboratory profile.
  Interventions: Drug: Anakinra

INTERVENTIONS:
Drug: Infliximab — Infliximab will be administered as a single IV dose of 10 mg/kg over 2 hours.
  Other Names: Remicade; Inflectra; Remsima
  Arms: Infliximab
Drug: Anakinra — Anakinra will be administered at a dose of 8 mg/kg/day IV or SQ with 100 mg every 6 hours as the max dose. This is discontinued with a taper during the hospitalization over 2-4 days once a patient is stable with significantly improved clinical course and laboratory profile.
  Other Names: Kineret
  Arms: Anakinra
Drug: Methylprednisolone — Methylprednisilone (steroids) will be administered as 2 mg/kg IV or orally divided every 12 hours. At the time of hospital discharge the patient will be given a steroid taper that will take at least 3 weeks to complete.
  Other Names: Steriods
  Arms: Methylprednisilone (steroids)

SUMMARY:
In March 2020, children exposed to the virus that causes the COVID-19 illness, SARS-CoV-2, presented with fever and significant inflammation about a month after exposure to the virus. Some children were sick enough to require care in the intensive care unit for what came to be known as Multisystem Inflammatory Syndrome-Children (MIS-C).The clinical presentation shared many features with Kawasaki disease (KD), a self-limited inflammation that can cause ballooning of the arteries of the heart. Thus, physicians reached for many of the therapies used to treat children with KD. Despite the surge of COVID-19 cases and children continuing to present with MIS-C, there are no data that guide the choice of therapy. Thus, the investigators have designed a study to determine which combination of therapies is most effective in helping children with MIS-C recover quickly.

DETAILED DESCRIPTION:
This study is a multi-site, randomized, pragmatic, comparative effectiveness study of children with MIS-C. The current standard of care is that all MIS-C patients are initially treated with IVIG and receive additional therapy if they are severely ill or do not improve clinically. This study design will randomize subjects who have received IVIG but clinically warrant further anti-inflammatory therapy to one of three treatment arms (infliximab, steroids or anakinra) and allow for re-randomization to one of the two remaining arms if clinically warranted.

ELIGIBILITY:
Inclusion Criteria:

1. An individual aged <21 years presenting with

   1. Fever (>38.0°C for ≥24 hours; may be by subjective report) AND
   2. Two or more of the following (from two different systems; e.g. one from cardiac and one from mucocutaneous):

      Cardiac
      * Hypotension
      * Shock
      * Arrhythmia
      * Tachycardia
      * Left ventricular ejection fraction <55%
      * Valvulitis
      * Coronary artery enlargement (LAD or RCA Z-score ≥ 2.5)
      * Pericardial effusion Gastrointestinal
      * Diarrhea
      * Nausea/vomiting
      * Significant abdominal pain Immunologic
      * Lymphadenopathy (unilateral cervical or diffuse) Mucocutaneous
      * Bilateral conjunctival injection
      * Extremity swelling or erythema
      * Rash
      * Lip erythema/Strawberry tongue Neurologic
      * Altered mental status
      * Focal neurological deficits
      * Headache
      * Meningismus
   3. Laboratory evidence of inflammation, including but not limited to, an elevated C-reactive protein (CRP), erythrocyte sedimentation rate (ESR), fibrinogen, procalcitonin, D-dimer, ferritin, lactic acid dehydrogenase (LDH), neutrophilia, lymphopenia or hypoalbuminemia AND
   4. No alternative plausible diagnoses based on clinical judgement AND
   5. Positive for current or recent SARS-CoV-2 infection by RT-PCR, serology, or antigen test; or suspected COVID-19 exposure AND
   6. Parent or legal guardian (or self if at least 18 years old) able and willing to provide informed consent and subject willing and able to provide assent when appropriate.

Exclusion Criteria:

1. Known immunodeficiency
2. Pre-existing medical condition that precludes receiving one or more of the study medications (e.g. TB, drug allergy to study medication).

Max Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 73 (Actual)
Dates: Start 2020-12-22 (Actual); Primary Completion 2023-12-22 (Actual); Study Completion 2024-04-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adriana Tremoulet, MD, MAS, Principal Investigator — University of California, San Diego
Locations (2):
- United States (2):
  - Rady Children's Hospital, San Diego, California
  - Children's Hospital Michigan, Detroit, Michigan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jain S, He F, Brown K, Burns JC, Tremoulet AH. Multisystem Inflammatory Syndrome therapies in children (MISTIC): A randomized trial. Contemp Clin Trials Commun. 2023 Apr;32:101060. doi: 10.1016/j.conctc.2023.101060. Epub 2023 Jan 20. PMID 36694613

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Infliximab | Methylprednisilone (steroids) | Anakinra
Started | 25 | 24 | 24
Completed | 25 | 24 | 22
Not Completed | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Infliximab | Methylprednisilone (steroids) | Anakinra | Total
Number analyzed (Participants) | 25 | 24 | 24 | 73
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 25 | 24 | 24 | 73
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 7.1 [4.76 to 12.6] | 7.95 [6.01 to 10.4] | 6.78 [4.95 to 9.6] | 7.64 [4.77 to 11.3]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 11 | 9 | 28
  Male | 17 | 13 | 15 | 45
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 2 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 5 | 1 | 4 | 10
  White | 15 | 20 | 19 | 54
  More than one race | 2 | 3 | 1 | 6
  Unknown or Not Reported | 1 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 25 | 24 | 24 | 73

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Needing Additional Anti-inflammatory Therapy Within the First Week of First Randomization
Description: The three arms of the study will be compared to see which initial randomization arm (infliximab, anakinra or steroids) has the lowest rate of additional anti-inflammatory therapy within the first week of first randomization.
Time Frame: 1 week
Measure: Count of Participants; unit: Participants
Arm/Group | Infliximab | Methylprednisilone (steroids) | Anakinra
Number analyzed (Participants) | 25 | 24 | 22
Participants | 10 | 10 | 14

2. Secondary Outcome: Number of Participants With Adverse Events
Description: Of the three initial randomization arms (infliximab, steroids or anakinra), the rate of adverse events will be compared. The goal is to determine which arm has the lowest rate of adverse events. The AEs reported in the AE section include: All Cause, SAE and Others.
Time Frame: 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Infliximab | Methylprednisilone (steroids) | Anakinra
Number analyzed (Participants) | 25 | 24 | 22
Participants | 0 | 16 | 1

ADVERSE EVENTS:
Time Frame: 6 weeks
Arm/Group | Infliximab | Methylprednisilone (steroids) | Anakinra
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/24 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/24 | 0/22
Other Adverse Events (participants affected / at risk) | 0/25 | 16/24 | 1/22
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Infliximab (N=25) | Methylprednisilone (steroids) (N=24) | Anakinra (N=22)
Bradycardia (Cardiac disorders) | 0 (0) | 9 (9) | 0 (0)
Hallucinations (Nervous system disorders) | 0 | 1 (1) | 1 (1)
Increased ALT (Hepatobiliary disorders) | 0 (0) | 2 (2) | 0 (0)
Melena (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Night Terrors (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
MRSA Skin Infection (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-13): https://cdn.clinicaltrials.gov/large-docs/31/NCT04898231/Prot_SAP_001.pdf